CLINICAL TRIAL: NCT05998980
Title: Clinical Comparison of Prefabricated Resin Composite Veneers and Direct Resin Composite Veneers Over 6-years
Brief Title: 6-year Clinical Performance of Prefabricated and Composite Veneers ( Componeer)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Sebnem Turkun, Prof. Dr, Ege University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16-2.1/8
Record Dates: First submitted 2023-08-11; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Dental Diseases; Tooth Discoloration
Keywords: veneers; prefabricated veneers; anterior restorations
MeSH Terms: conditions — Stomatognathic Diseases; Tooth Discoloration

STUDY DESIGN:
Intervention Model Description: Individual Randomized Assignment
Who Masked: Participant, Care Provider
Masking Description: Double (Participant, Evaluator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Componeer Prefabricated Veneers (Active Comparator): Componeer veneers (device 1) were randomly applied to patients. The teeth were evaluated in terms of color and size matching in order to select the correct veneers. Componeer sizing guide was used for size selection. Prefabricated veneers were adapted to the teeth' surfaces. Then, the inner surfaces of the prefabricated veneers were roughened to obtain better mechanical retention. Then the labial surfaces of the teeth were etched using 36% phosphoric acid. The etched surfaces were rinsed and dried. An adhesive system was applied to the teeth. Prefabricated veneers' inner surfaces were cleaned with alcohol, and One Coat dental adhesive was applied. Synergy D6 nanohybrid resin composite was placed on the inner surfaces of the veneers and transferred to the teeth. The restorations were light-cured for 40 s Gingival borders were adapted with contouring and polishing discs (intervention 1).
  Interventions: Procedure: Componeer prefabricated veneers
- Essentia resin composite venners (Active Comparator): Direct resin composite restorations were randomly applied to patients. Essentia resin composite (device 2) shade guide was used for color selection. After the preparation, the labial surfaces of the teeth were etched using 36% phosphoric acid. The etched surfaces were then rinsed and dried. An adhesive system G-Premio Bond was applied to the teeth. Then Essentia micro-hybrid resin composite with dentin shade was placed on labial surfaces of teeth and was light-cured. Then enamel shade was placed on the tooth. After that, the resin composite veneer was light-cured for 20 s from each surface. Proximal surfaces were polished using proximal sandpaper strips (intervention 2).
  Interventions: Procedure: Essentia resin composite veneers

INTERVENTIONS:
Procedure: Componeer prefabricated veneers — Individual Randomized Clinical Trial
  Arms: Componeer Prefabricated Veneers
Procedure: Essentia resin composite veneers — Individual Randomized Clinical Trial
  Arms: Essentia resin composite venners

SUMMARY:
The aim of this study is to compare the clinical performance of composite veneers performed in two different ways, indirect and direct methods over a period of 6-year.

30 volunteer patients without systemic diseases and who applied to Ege University School of Dentistry for the esthetic restoration of their anterior diastema (gap) were selected according to inclusion and exclusion criteria. The closure of 102 diastema was randomly performed with prefabricated composite resin veneers (n=15; indirect method- Componeer, Coltène, Altstätten, Switzerland) or direct composite resin veneers (n=15; direct method- Essentia, GC, Japan). These restorations were clinically evaluated at baseline, 1-2-6-year by two experienced and blind examiners according to modified Ryge criteria (USPHS criteria). Color match, marginal discoloration, anatomic form, marginal adaptation, secondary caries, surface roughness, retention, and polishing retention were evaluated for that purpose. Statistical analysis was performed with McNemar and Chi-square tests (p<0.05).

DETAILED DESCRIPTION:
The aim of this study is to compare the clinical performance of composite veneers performed in two different ways, indirect (Componeer) and direct methods (Essentia) over a period of 6-year.

The study protocol was approved by the Ethical Committee of Ege University, Izmir, Turkey (16-2.1/8; 01.04.2016). 30 patients without any systemic diseases (10 males, 20 females, mean age: 34) and with aesthetic complaints on their anterior teeth were treated with 102 restorations (48 Componeer and 54 Essentia).

In Group 1; 48 teeth (15 patients) were restored with Componeer prefabricated veneers (Coltène, Altstätten, Switzerland) in combination with Synergy D6 nanohybrid resin composite (Coltène) and One Coat Bond (Coltène) adhesive system. In Group 2; 54 teeth (15 patients) were restored with Essentia (GC, Japan) micro-hybrid resin composite in combination with G-Premio Bond (GC) adhesive system.

Periodontal treatments, fillings, and bleaching treatments were performed, if necessary, before any veneer treatment. For the pre-treatment records; 3 photographs (smile, anterior occlusion, and upper anterior teeth alone) were taken from each patient. Both groups used the "Button Try" technique for color selection. Componeer sizing guide was used for size selection in Group 1. Then teeth were cleaned with non-fluoride pumice (Cleanic; Kerr Dental, ABD) using a polishing brush. Isolation of the teeth and retraction of the lips were achieved with a rubber dam (OptraDam, Ivoclar Vivadent, Liechtenstein). Prefabricated veneers were prepared for the cementation process in Group 1. Then the labial surfaces were etched using 36% phosphoric acid for 30 s. The etched surfaces were rinsed for 30 s and dried. One Coat Bond (Coltene) adhesive system was applied on the labial surfaces of the teeth in accordance with user instructions in both groups. In Group 1; Synergy D6 nano hybrid resin composite was placed on the inner surfaces of the prefabricated veneers before being applied on appropriate teeth. Then the restorations were light-cured for 40 s from each surface (D-Light Pro, GC) and polished with a polishing paste (Prisma Gloss Extra Fine, Dentsply, NY, ABD) and a felt wheel.

In Group 2; Essentia (GC) micro-hybrid resin composite with dentin color was placed on the labial surfaces of the teeth and light-cured (D-Light Pro, GC). After that layer, Essentia enamel shades were placed over the labial surface of the tooth and light-cured for 20 s from each surface. The diamond bur contouring was performed and polishing discs (Super-Snap Rainbow Technique Kit, SHOFU) were used. For polishing purposes, a polishing paste (Prisma Gloss Extra Fine, Dentsply, NY, ABD) and a felt Wheel were used.

In group 1; gingival borders were adapted with contouring and polishing discs (Super-Snap Rainbow Technique Kit, SHOFU). Then proximal surfaces were polished using proximal sandpaper strips. Occlusion was checked for premature contacts. Two calibrated observers who were blinded to the objective of this study performed the evaluations. Color match, marginal adaptation, marginal discoloration, anatomic form, retention, secondary caries, and gloss retention were the properties evaluated for the restorations at baseline, 1-2-6-year using Modified Ryge Criteria (USPHS Criteria). Statistical analysis was performed with McNemar and Chi-square tests (p<0.05).

ELIGIBILITY:
Inclusion Criteria:

* Being healthy without any chronic disease
* Having diastema in the anterior teeth without any caries
* Not having an occlusal anomaly such as bruxism or anterior crossbite
* Having a good oral hygiene
* Agreeing to come to the recall sessions regularly for 6 years
* Being over the age of 18

Exclusion Criteria:

Exclusion Criteria:

* Having uncontrolled parafunction such as bruxism or anterior deep bite
* Having insufficient oral hygiene
* Being pregnant
* Having a systemic disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2017-01-15 (Actual)

PRIMARY OUTCOMES:
Marginal discoloration | 6 years
  Marginal discoloration of prefabricated and resin composite veneers Evaluating differently veneer options on anterior teeth with United State Public Health Service criteria regarding marginal discoloration by 2 independent evaluators Marginal discolouration was evaluated by 2 independent clinicians. Visual inspection with a mirror at 18 inches was performed. A score means the higher score of clinical acceptability while C score means that the restoration has failed and needs to be replaced.
  Alpha: No discoloration anywhere along the margin between the restoration and the adjacent tooth. Bravo: Slight discoloration along the margin between the restoration and the adjacent tooth.
  Charlie: The discoloration penetrated along the margin of the restorative material in a pulpal direction.
Marginal adaptation | 6 years
  Marginal adaptation of prefabricated and resin composite veneers Evaluating differently veneer options on anterior teeth with United State Public Health Service criteria regarding marginal adaptation by 2 independent evaluators Marginal discolouration was evaluated by 2 independent clinicians. Visual inspection with a mirror at 18 inches was performed . A score means the higher score of clinical acceptability while C score means that the restoration has failed and needs to be replaced.
  Alpha: No discoloration anywhere along the margin between the restoration and the adjacent tooth. Bravo: Slight discoloration along the margin between the restoration and the adjacent tooth.
  Charlie: The discoloration penetrated along the margin of the restorative material in a pulpal direction.
Retention rate | 6 years
  Retention rates of prefabricated and resin composite veneers Evaluating differently veneer options on anterior teeth with United State Public Health Service criteria regarding retention rates by 2 independent evaluators Marginal discolouration was evaluated by 2 independent clinicians. Visual inspection with a mirror at 18 inches was performed . A score means the higher score of clinical acceptability while C score means that the restoration has failed and needs to be replaced.
  Alpha: No discoloration anywhere along the margin between the restoration and the adjacent tooth. Bravo: Slight discoloration along the margin between the restoration and the adjacent tooth.
  Charlie: The discoloration penetrated along the margin of the restorative material in a pulpal direction.
Anatomic form | 6 years
  Anatomic form of prefabricated and resin composite veneers Evaluating differently veneer options on anterior teeth with United State Public Health Service criteria regarding anatomic form by 2 independent evaluators Marginal discolouration was evaluated by 2 independent clinicians. Visual inspection with a mirror at 18 inches was performed. A score means the higher score of clinical acceptability while C score means that the restoration has failed and needs to be replaced.
  Alpha: No discoloration anywhere along the margin between the restoration and the adjacent tooth. Bravo: Slight discoloration along the margin between the restoration and the adjacent tooth.
  Charlie: The discoloration penetrated along the margin of the restorative material in a pulpal direction.
Color match | 6 years
  Color changes of prefabricated and resin composite veneers Health Service criteria regarding color changes by 2 independent evaluators Marginal discolouration was evaluated by 2 independent clinicians. Visual inspection with a mirror at 18 inches was performed . A score means the higher score of clinical acceptability while C score means that the restoration has failed and needs to be replaced.
  Alpha: No discoloration anywhere along the margin between the restoration and the adjacent tooth. Bravo: Slight discoloration along the margin between the restoration and the adjacent tooth.
  Charlie: The discoloration penetrated along the margin of the restorative material in a pulpal direction

CONTACTS AND LOCATIONS:
Overall Officials: Sebnem L Turkun, DDS,PhD, Study Director — Ege University
Locations (1):
- Ege University School of Dentistry Department of Restorative, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No